CLINICAL TRIAL: NCT06066138
Title: A Feasibility Phase I Study of Therapeutic Drug Monitoring-Based Atezolizumab Dosing
Brief Title: A Study of Therapeutic Drug Monitoring-Based Atezolizumab Dosing
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001559; 001559-C
Record Dates: First submitted 2023-10-03; First posted 2023-10-04 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12-16

CONDITIONS: Locally Advanced Alveolar Soft Part Sarcoma; Metastatic Alveolar Soft Part Sarcoma; Locally Advanced Non Small Cell Lung Cancer; Metastatic Non Small Cell Lung Cancer; Locally Advanced Small Cell Lung Cancer; Metastatic Small Cell Lung Cancer; Locally Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma; Locally Advanced Melanoma; Metastatic Melanoma
Keywords: PD-L1; PD-1; Tecentriq; Immunotherapy
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular; Melanoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Atezolizumab treatment course
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab administered via IV at either 1,200 mg q3 weeks, or 1,680 mg q4 weeks for the first 2 doses followed by 840mg q2 weeks or q6 weeks.

SUMMARY:
Background:

A type of drug called monoclonal antibody immune checkpoint inhibitors are often used in cancer treatment. These drugs help the body s immune system fight cancer by blocking proteins that cause cancer cells to grow. One of these drugs (atezolizumab) is approved to treat certain cancers. Researchers want to find out if lower doses of this drug might provide the same benefit with fewer adverse effects.

Objective:

To test different doses and timing of atezolizumab for people with cancer.

Eligibility:

People aged 18 years and older with cancer that has spread locally or to other organs. They must be eligible for treatment with the study drug.

Design:

Participants will be screened. They will have blood tests and imaging scans. They will provide a sample of tissue from their tumor.

Atezolizumab is administered through a tube attached to a needle inserted into a vein in the arm. Participants will take this drug alone or combined with other drugs prescribed for their care.

The first 2 treatments will be done per the FDA recommended dose and schedule. Before administering the second dose of the study drug, researchers will check the level of the drug in the participant s blood. Depending on those results, their 3rd dose will be scheduled 2 to 6 weeks later.

For the 3rd dose of the study drug, participants will switch to the FDA minimum dosage. Dosages of any other drugs will not change.

Researchers will continue to test the levels of the drug in participants blood before each treatment for 16 weeks. After that, these levels will be tested every 3 months.

Study treatment may last up to 2 years.

DETAILED DESCRIPTION:
Background:

* The treatment of many cancers has been revolutionized through the use of monoclonal antibody immune checkpoint inhibitor drugs, particularly those that block the interaction of the anti-programmed death-ligand 1 (PD-L1) with the programmed death-1 (PD-1) receptor.
* Atezolizumab was initially tested in a phase 1a multicenter, dose-escalation, and dose- expansion study (NCT01375842) which showed that the drug was well tolerated and produced clinical responses in a variety of tumors.
* The initially approved atezolizumab regimen was 1,200 mg every 3 weeks, but 840 mg every 2 weeks was added based on the data from the TNBC trial (NCT01375842). This was taken further by Morrissey et al., who used population pharmacokinetic (PK) simulations to determine that dosing regimens of 840 mg every 2 weeks and 1,680 mg every 4 weeks are interchangeable with 1,200 every 3 weeks in terms of efficacy, leading the Food and Drug Administration (FDA) to expand the dosing regimens for atezolizumab.
* The standard dosing regimens yield steady-state concentrations greater than 10-fold above the stated minimum effective concentration of 6 microg/mL, to ensure adequate exposure for all patients, including patients that may experience lower exposure due to the incidence of anti-drug-antibodies (ADA). Atezolizumab exhibits a flat exposure- response relationship.

Objective:

-To test the feasibility of reducing drug exposure while maintaining plasma drug concentration at or above the expected target trough value during a 16-week study period by using a method for therapeutic drug monitoring of atezolizumab.

Eligibility:

* Age >= 18 years old.
* Participants with a locally advanced or metastatic cancer whose NCI Licensed Independent Practitioner (LIP) determined they are candidates for treatment with atezolizumab, either alone or in combination with other FDA-approved drug(s).
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
* Adequate organ and marrow function.

Design:

* This is a phase I feasibility study of a therapeutic drug monitoring (TDM)-based method for atezolizumab dosing.
* The participants will start with FDA approved dose and frequency of atezolizumab (840 mg every 2 weeks, 1,200 mg every 3 weeks, or 1,680 mg every 4 weeks) selected by their treating physician for the first two doses of the drug per standard of care.
* After the second dose, starting at 3rd dose, the dose of the drug will be switched to 840 mg and will be used going forward in the trial in all participants.
* Prior to each dose a trough will be drawn which will be by the population PK model to predict the timing of the next dose to maintain the atezolizumab target trough for each

participant specifically. This will be repeated for the first 16 weeks of treatment.

-After 16 weeks of treatment, the timing of the next dose to maintain the atezolizumab target trough for each participant will be monitored and adjusted (if necessary) every 3 months for each participant until 2 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants with a locally advanced or metastatic pathologically confirmed cancer whose NCI Licensed Independent Practitioner (LIP) determined they are candidates for treatment with atezolizumab, either alone or in combination with other FDA-approved drug(s), for example, TMB-high, PDL-1 positive, or other disease states that respond to PD(L)-1 inhibitors. Regimens with atezolizumab alone or in combination with agents that have previously demonstrated safety in published clinical trials may be used. An LIP may be either an MD, DO, PA, or NP and must be qualified for oncologic management per institutional practice.
* Age >=18 years old.
* Measurable disease per RECIST 1.1 criteria.
* ECOG performance status of 0-2.
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) >=1,200/microliter
  * Hemoglobin >9.0 g/dL
  * Platelets >=75,000/microliter
  * Total bilirubin <= 1.5 mg/dL, except in participants with Gilbert s Syndrome who must have a total bilirubin less than 3.0 mg/dL
  * Aspartate aminotransferase (AST) / Alanine aminotransferase (ALT) <=2.5 X institutional upper limit of normal (ULN)
  * Creatinine Clearance (CrCl) >=30 mL/min/1.73 m^2 (calculated using the Cockcroft-Gault formula).
  * Serum albumin > 3 g/dL
* Individuals of child-bearing potential (IOCBP) must agree to use a highly effective method of contraception (hormonal, intrauterine device (IUD), surgical sterilization) for the duration of the study treatment and up to 5 months after the last dose of the atezolizumab (restriction period). NOTE: abstinence, defined as no vaginal heterosexual intercourse within 6 months prior to the treatment initiation and willingness to continue abstinence for restriction period is also acceptable.

Individuals who can father children must agree to use an effective method of contraception (barrier, surgical sterilization) at study entry and up to 5 months after the last dose of the atezolizumab.

* Nursing participants must be willing to discontinue nursing from study treatment initiation through 5 months after atezolizumab treatment discontinuation.
* Participants with history of human immunodeficiency virus (HIV) infection must be on effective anti-retroviral therapy and have undetectable viral load.
* Participants with history of chronic hepatitis B virus (HBV) infection must be on suppressive therapy, if indicated, and have undetectable HBV viral load.
* Participants with history of hepatitis C virus (HCV) infection must have an undetectable HCV viral load.
* Participants with history of treated brain metastases must have follow-up brain imaging after central nervous system (CNS)-directed therapy with no evidence of progression.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible.
* All participants must have the ability to understand and willingness to sign a written informed consent.

EXCLUSION CRITERIA:

Participants who have received an investigational agent for treating participants' disease not approved by FDA within 28 days prior to study treatment initiation.

* Participants who have received immunostimulatory agents, including, but not limited to, IFN-alpha, IFN-gamma, or IL-2, immunosuppressive medications, and any herbal medicines within 1 month prior to study treatment initiation. NOTE: Physiologic doses of systemic steroids (<= 10 mg prednisone or equivalent) or local (e.g., topical, nasal, intraarticular, inhaled) steroid use is permitted.
* Prior treatment with CD137 agonists
* Prior treatment with immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies; (including atezolizumab) within 28 days prior to study treatment initiation.
* History or risk of autoimmune disease, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone.
  * Participants with controlled Type 1 diabetes mellitus on a stable insulin regimen.
  * Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis would be excluded) are permitted provided all of the following conditions are met:

    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at screening and only requiring low potency topical steroids
    * No acute exacerbations of underlying condition within 12 months prior to study treatment initiation (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids) within 12 months prior to study treatment initiation.
* Persisting toxicity related to prior therapy of Grade >1 per Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 unless deemed not clinically significant or irreversible. NOTE: alopecia and sensory neuropathy Grade <= 2 are acceptable.
* Participants with prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment
* Active tuberculosis at screening
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Participants with significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident (https://www.heart.org/en/health-topics/heart-failure/what-isheart-failure/classes-of-heart-failure), unstable arrhythmia, or unstable angina within 3 months prior to study treatment initiation.
* Pregnancy (confirmed with Beta-Human chorionic gonadotropin (Beta-HCG) serum or urine pregnancy test in IOCBP performed at screening).
* Uncontrolled intercurrent illness or situation that would limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of reducing drug exposure while maintaining plasma drug concentration | 16 weeks
  The fraction of participants that can be dosed with 840mg of atezolizumab at less frequent intervals while maintaining a trough PK concentration at or above 6 mg/mL

SECONDARY OUTCOMES:
Minimal frequency (median, range) of atezolizumab dosing to keep the trough concentration at or above 6 microgram/mL | 16 weeks and every 3 months on treatment
  PK evaluations before every atezolizumab infusion starting from the second dose until 16 weeks after atezolizumab treatment and every 3 months after 16 weeks on treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers within 10 years after the completion of the primary endpoint by contacting the NCI Principal Investigator.
Access Criteria: Data from this study may be requested by contacting the NCI Principal Investigator

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001559-C.html